CLINICAL TRIAL: NCT06825234
Title: Prognostic Value of a Multidimensional Assessment for Survival in Elderly Patients With CKD 4B/5
Acronym: PROFILER
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/912
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease Stage 5; Chronic Kidney Disease Stage 4B
Keywords: Frailty; Patient-Related Outcomes; Personalised care
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine a multidimensional signature (integrating frailty and patient-reported outcomes measures (PROMs) at entry into stage 4B/5 CKD) to improve prediction of renal death (dialysis, transplantation, conservative management, death).

DETAILED DESCRIPTION:
In 2019, 4,263 patients starting dialysis in France were aged 75 years or older. This elderly population, often with comorbidities, poses a number of challenges for nephrologists, both in terms of initiation and modalities of dialysis and access to transplantation. Dialysis may offer little benefit in terms of survival, often at the cost of a significant impact on quality of life and number of hospitalisations. There is a current trend to offer conservative treatment as an alternative to dialysis. However, there are no objective criteria to guide this decision and the uremic syndrome may distort certain clinical perceptions. The aim of this study is to determine whether an assessment that incorporates multiple dimensions, including those of frailty, can help the clinician determine the best course of treatment for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stage 4B or 5 (first consultation with GFR < 20 mL/min /1.73 m2 in CKD-EPI 2009).
* Fluency in French
* Membership of a French social security scheme
* Non-opposition from the subject to participate in the study

Exclusion Criteria:

* Subjects with limited legal capacity.
* Subjects still in the exclusion period of another study, or according to the national registry of clinical trial participants.
* Subjects with no social security coverage.
* Subjects judged by the investigator to be unlikely to comply with study procedures
* Subjects unable to understand the reasons for the study; psychiatric disorders judged by the investigator to be incompatible with inclusion in the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population consisted of patients aged 75 years and older with stage 4B/5 chronic kidney disease (GFR<20ml/min/1.73m²), who spoke French and were under the usual care of the nephrology units involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  Time between first visit (entry into stage 4B/5) and death from any cause. Living patients will be censored at the date of last news. Entry into CKD 4B/5 is defined as the first kidney disease follow-up visit for which the patient has an eGFR strictly below 20 ml/min/1.73m2.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Besançon University Hospital, Besançon
  - Tours University Hospital, Tours